CLINICAL TRIAL: NCT01301105
Title: The Effects of Mindfulness Training on Pain Regulation, Negative Affect, Attention, and Social Stress.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AT002114-01
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-05

CONDITIONS: Focus on Pain Regulation Mechanisms; Social Stress Mechanisms; Basic Affective Mechanisms; Attention Mechanisms; Brain Mechanisms; Immune Mechanisms; Endocrine Mechanisms
Keywords: pain regulation; social stress; affect; attention; brain; immune; endocrine
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Enhancement Program (HEP) (Placebo Comparator): Intervention designed to be effective and structurally equivalent to Mindfulness Based Stress Reduction (MBSR) but without a mindfulness component. Designed as an active control for MBSR to isolate mindfulness as an active ingredient.
  Interventions: Behavioral: Health Enhancement Program (HEP)
- Mindfulness Based Stress Reduction (MBSR) (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — 8 week class in stress reduction through instruction in mindfulness related techniques.
  Arms: Mindfulness Based Stress Reduction (MBSR)
Behavioral: Health Enhancement Program (HEP) — 8-week intervention designed to be structurally equivalent to MBSR but without a mindfulness component. Consists of nutrition, functional movement, physical activity, and music therapy.
  Arms: Health Enhancement Program (HEP)

SUMMARY:
The project's objective is to explore the impact of Mindfulness-Based-Stress-Reduction (MBSR) on pain regulation, social stress, basic affective and attention functions, and on the brain, immune, and endocrine mechanisms that subserve these processes. Specifically, the investigators hypothesize that participants undergoing MBSR training will show decreased emotional distress on self-report measures, increased sustained attention on a behavioral task, decreased stress levels on a social stress test, decreased general psychosocial stress as indexed by diurnal salivary cortisol profile, changes in inflammatory response, modulation of cellular aging, and different neural patterns in response to thermal pain and aversive visual stimuli as indexed by functional Magnetic Resonance Imaging (fMRI).

To test these hypotheses, the study will recruit 50 participants through the UW-Madison Integrative Medicine Program. All participants will be randomly assigned either to an 8-week MBSR program or to an 8-week training program in health-enhancement. At the conclusion of the study, participants will be invited to participate to the second class should they be interested. Participants will complete self-report questionnaires, behavioral tasks, fMRI scanning, cortisol sampling, and blood sampling before training begins, after the first program ends, and again four months after the first program ends and prior to the second program.

If hypotheses are supported, the study may benefit participants by reducing their psychological distress, increasing their well-being, and helping them better manage pain and aversive stimuli. There are no other direct benefits to participants. Potential risks associated with fMRI include ferromagnetic collision, neurostimulation effects, and psychological discomfort. Potential risks to subjects include slight potential discomfort in providing saliva samples, discomfort of painful thermal stimulation, stress associated with the Trier Social Stress Test, some psychological discomfort from viewing disturbing photographs as part of the compassion fMRI study, and breach of confidentiality.

Consent for the present study will entail both written and verbal descriptions of the protocol. Subjects will be informed that their participation is completely voluntary, and that they can withdraw at any time.

ELIGIBILITY:
Inclusion Criteria:

1.1 Risk Factors

* Able to lie still in the scanner for 90 minutes
* Weighs under 300 pounds

1.2 Factors impacting on the outcome measures

* 18-65 years old
* Right-handed
* No previous experience with meditation.
* No daily practice with other mind-body techniques (e.g., yoga, tai-chi, but previous exposure to yoga is okay)
* In good general health as determined by the investigator

1.3 Logistic Issues

* Able to walk
* Able to understand and speak English
* Able to provide written consent prior to admission
* Able to see without glasses (as if looking through binoculars)

Exclusion Criteria:

2.1 Risk Factors

* Any metallic implants, such as prostheses that cannot be removed, aneurysm clip-S, dental or orthodontic (filings are okay), or orthopedic (e.g., pins, rods, screws, nails) [okay with doctors note]
* Any electronic implants, such as cardiac pacemakers, cardiac defibrillator, artificial heart valve, cardiac pace wires,
* Lens implants prior to 1983
* Breast/penile, electrodes, neurostimulators/biostimulators, pumps (e.g. drug infusion device), bone or socket implants (Check with PI or MR technician)
* Any type of prosthesis
* Any permanent cosmetics (e.g., eyeliner) prior to 1975
* Any tattoos on upper body prior to 1975
* Any irremovable non plastic body piercing(s)
* Has ever worked as an occupational metal grinder without protective glasses
* Has ever worked with metal as a hobby without protective glasses
* Has ever had or sought medical attention for metal in the eyes [requires orbit x-ray]
* Has ever has metal fragments removed from eyes [requires orbit x-ray]
* Has ever been struck by a gun shot, B.B. or shrapnel, and the bullet stuck [judgement]
* Has a history of any metal in body
* Diabetes
* Peripheral vascular disease, peripheral arterial disease, Raynaud's disease, or any other diagnosed circulatory disorders
* Body mass index (BMI) below 18.5
* Any involuntary motor disorders
* Has a cochlear implant
* Wears a hearing aid that cannot be taken out (Check with PI or MR technician)
* Wears a hearing aid
* Wears dentures that cannot be removed or contain metal
* A subject who is claustrophobic
* A female subject who is pregnant or has an intrauterine device (IUD)
* Allergic to adhesive tape
* A history of problems of any kind during blood draws
* Women who may be pregnant
* Women who have an intrauterine device (IUD) [okay with a doctors note]
* 2 or more of the following [judgment]
* Diagnosed hypertension?
* Hyperlipidemia
* High cholesterol
* Obesity can be calculated from weight & height info.
* Smoke cigarettes
* Family history of coronary or atherosclerotic disease (parents/siblings prior to age 55)

2.2 Factors impacting on the outcome measures

* Current medical disorders that might make interpretation of scan data difficult
* Has a problem with alcohol or non prescription drugs
* Use of medications that affects CNS function, including psychotropics, opiate medication or corticosteroids, during the last 3 months
* Any prescribed psychotropic medications, currently or during the last 3 months (These include medications for anxiety, depression, or other psychological problems)
* Plans to start taking any prescribed psychotropic medications
* Takes inhaled steroids for asthma? (e.g., Fluticasone)
* Takes any corticosteroids?
* Night shift workers (11 pm to 7 am) d/t potential disruption of cortisol level variability
* Diabetes requiring insulin treatment
* Has TMJ (Temporal Mandibular Joint) disorder or other problems with biting/chewing
* Previous training in meditation
* Currently meditates on a regular basis
* Daily yoga, tai-chi, or Qigong practice
* Engagement in moderate sport and recreational activities more than 5 times a week
* Engagement in vigorous sport and recreational activities more than 4 times a week

2.3 Logistic Issues

* Phobia of needles
* Not able to attend an informational session, all class meetings, and all clinic visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Lutz, Ph.D., Principal Investigator — UW-Madison; Richard Davidson, Ph.D., Study Director — UW-Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] MacCoon DG, MacLean KA, Davidson RJ, Saron CD, Lutz A. No sustained attention differences in a longitudinal randomized trial comparing mindfulness based stress reduction versus active control. PLoS One. 2014 Jun 23;9(6):e97551. doi: 10.1371/journal.pone.0097551. eCollection 2014. PMID 24955584